CLINICAL TRIAL: NCT00402714
Title: A Randomized Trial of Extracorporeal Photopheresis, Pentostatin, and Total Body Irradiation Versus Pentostatin and Total Body Irradiation in Patients Undergoing Reduced Intensity Allogeneic Stem Cell Transplantation for the Treatment of Malignancies
Brief Title: A Trial of Extracorporeal Photopheresis, Pentostatin, and Total Body Irradiation in Patients Undergoing Reduced Intensity Allogeneic Stem Cell Transplantation for the Treatment of Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0508000433
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Hematologic Malignancies
Keywords: Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Photopheresis; Methoxsalen; Pentostatin; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Extracorporeal photopheresis, pentostatin and total body irradiation
  Interventions: Procedure: extracorporeal photopheresis; Drug: Pentostatin; Radiation: Total Body Irradiation
- 2 (Active Comparator): Pentostatin and total body irradiation
  Interventions: Drug: Pentostatin; Radiation: Total Body Irradiation

INTERVENTIONS:
Procedure: extracorporeal photopheresis — Extracorporeal photopheresis (ECP) is the ex vivo exposure of the leukocyte rich fraction to ultraviolet light in the presence of 8-methoxypsoralen.
  Other Names: UVAR® XTS Photopheresis System; UVADEX®; 8-methoxypsoralen; methoxsalen
  Arms: 1
Drug: Pentostatin — pentostatin 8mg/m2 over 48 hours by continuous infusion
  Other Names: DCF; 2-Deoxycoformycin; Nipent
  Arms: 1
Radiation: Total Body Irradiation — 600cGy TBI in 3 200cGy TBI fractions
  Arms: 1
Drug: Pentostatin — pentostatin 8mg/m2 over 48 hours by continuous infusion
  Other Names: DCF; 2-Deoxycoformycin; Nipent
  Arms: 2
Radiation: Total Body Irradiation — 600cGy TBI in 3 200cGy TBI fractions
  Arms: 2

SUMMARY:
This is a study to explore the use of a reduced intensity transplant conditioning regimen. A conditioning regimen is the treatment that is given to prepare a body for the new bone marrow that will be received from a donor. Reduced intensity conditioning uses lower doses of chemotherapy than conventional conditioning regimens. The use of lower doses of drugs and radiation cause fewer side effects. Reduced intensity regimens have been offered to older patients or patients at increased risk for transplant-related side effects and have been shown to be safe and effective. Reduced intensity conditioning regimens are now considered for many patients who are undergoing transplant.

DETAILED DESCRIPTION:
One of the complications of allogeneic stem cell transplant (ASCT) is graft versus host disease (GVHD). This is when the donor cells that are infused attack the body organs. This can cause serious illness and even death. The chance of getting serious life threatening GVHD with conventional transplant conditioning regimens is 25-50% depending on whether the donor bone marrow is from a family member or an unrelated person. The reduced intensity conditioning regimen used in this study involves a drug called pentostatin as well as a reduced dose of radiation and a treatment called photopheresis. This regimen has been successfully used in 106 patients. The incidence of serious GVHD in those patients was much less than expected: 8% for patients getting bone marrow from a family member and 23% for those getting bone marrow from an unrelated person. The pentostatin and radiation parts of this reduced intensity conditioning regimen are similar to other types of reduced intensity regimens, which use drugs similar to pentostatin. The unique part of this regimen compared to others is the use of extracorporeal photopheresis (ECP).

While ECP has been used in 106 patients as part of a reduced intensity conditioning regimen, it is unknown whether adding ECP to pentostatin and radiation is what caused the reduced rate of GVHD that was seen in the previous study that was done. The use of ECP as part of a conditioning regimen is investigational. ECP is approved by the U.S. Food and Drug Administration (FDA) for the treatment of cutaneous T-cell lymphoma, but is not approved by the FDA for use prior to ASCT.

Because it is not known whether the use of ECP in the reduced intensity conditioning regimen was what caused the low incidence of GVHD, this research study will look at differences in getting GVHD based on whether you receive ECP. Half the patients in this research study will receive ECP as part of their reduced intensity-conditioning regimen and the other half will not. Patients will be randomized (50% chance you will receive ECP and 50% chance you will not). Both groups will receive pentostatin and reduced dose total body irradiation. The primary purpose of this research study is to look at the chance of developing serious GVHD within the first 100 days after transplant within each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give informed consent to receive study treatment.
* Availability of a suitable 5/6 (Class I mismatch) or 6/6 HLA-matched related or 10 or 10 matched unrelated donor.
* Adequate cardiac function with an ejection fraction ≥ 35% by echocardiography or nuclear cardiography within three months of transplantation
* Adequate pulmonary function with corrected DLCO ≥ 40% by pulmonary function testing within the past three months of transplantation
* Adequate renal function with creatinine clearance ≥ 30 ml/min. as calculated by the Cockroft and Gault method.
* Adequate hepatic function with AST, ALT, alkaline phosphatase, and total bilirubin no more than 3 x ULN unless related to neoplastic disease.
* Adequate vascular access, either by pheresis flow catheter or peripheral vein intravenous catheter, to perform ECP, should the patient be randomized to ECP.
* Patients with prior autologous stem cell transplantation are eligible.
* Age 18 to 75 years.
* Life expectancy of greater than 3 months.
* ECOG performance status of 0, 1, or 2.
* Platelet counts ≥ 20,000/microliter, with or without transfusion support, at the time of ECP, should the patient be randomized to ECP.
* Weight ≥ 40 kg.
* Systolic blood pressure ≥ 90 mmHg on the day randomization occurs
* Negative pregnancy test. The effects of ECP on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Able to receive 600 cGy of total body irradiation. If patient previously treated by TBI then must be able to receive 400cGY of total body irradiation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Hypersensitivity or allergy to 8-methoxypsoralen.
* Prior allogeneic stem cell transplantation
* HLA-DR mismatch or no worse than one antigen-mismatched unrelated donor.
* Patients with acute leukemia or acute lymphocytic leukemia with > 5% circulating blasts in peripheral blood or > 5% blasts in bone marrow aspirate and biopsy at the time of registration
* Patients with chemorefractory non-Hodgkin's lymphoma or Hodgkin's disease or multiple myeloma
* Diagnosis of myelofibrosis
* Patients known to be positive for antibodies to HIC or have evidence for active HIC viral replication.
* Participation in another clinical trial for prevention of GVHD.
* Patient is pregnant or lactating.
* Lack adequate vascular access for ECP.
* Systolic blood pressure < 90 mmHg at the time of randomization, should the patient be randomized to ECP.
* Evidence of active, ongoing infection.
* Unwilling to comply with all study procedures.
* Unable or unwilling to give signed informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, M.D., Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Methodist Hospital - Texas Transplant Institute, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ECP/Pent: Extracorporeal photopheresis, pentostatin and total body irradiation
  extracorporeal photopheresis: Extracorporeal photopheresis (ECP) is the ex vivo exposure of the leukocyte rich fraction to ultraviolet light in the presence of 8-methoxypsoralen.
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
- Pent: Pentostatin and total body irradiation
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
Period: Overall Study
Arm/Group | ECP/Pent | Pent
Started | 3 | 11
Completed | 3 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pent/TBI
Groups:
- 1 ECP and Pent/TBI: Extracorporeal photopheresis, pentostatin and total body irradiation
  extracorporeal photopheresis: Extracorporeal photopheresis (ECP) is the ex vivo exposure of the leukocyte rich fraction to ultraviolet light in the presence of 8-methoxypsoralen.
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
- 2 Pent/TBI: Pentostatin and total body irradiation
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
- Total: Total of all reporting groups
Arm/Group | 1 ECP and Pent/TBI | 2 Pent/TBI | Total
Number analyzed (Participants) | 3 | 11 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 0 | 3 | 3
Gender [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 2-4 Acute Graft Versus Host Disease Following Allogeneic Stem Cell Transplantation in Patients Randomized to Photopheresis vs. no Photopheresis
Time Frame: Day +100 following allogeneic stem cell transplant
Measure: Number; unit: participants
Arm/Group | 1 ECP and Pent/TBI | 2 Pent/TBI
Number analyzed (Participants) | 3 | 11
participants | 1 | 8

2. Secondary Outcome: Overall Survival
Time Frame: 2 years following stem cell transplant
Measure: Number; unit: participants
Groups:
- ECP Pento TBI: Extracorporeal photopheresis, pentostatin and total body irradiation
  extracorporeal photopheresis: Extracorporeal photopheresis (ECP) is the ex vivo exposure of the leukocyte rich fraction to ultraviolet light in the presence of 8-methoxypsoralen.
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
- Pento TBI: Pentostatin and total body irradiation
  Pentostatin: pentostatin 8mg/m2 over 48 hours by continuous infusion
  Total Body Irradiation: 600cGy TBI in 3 200cGy TBI fractions
Arm/Group | ECP Pento TBI | Pento TBI
Number analyzed (Participants) | 3 | 11
participants | 2 | 5

ADVERSE EVENTS:
Arm/Group | ECP/Pent | Pent
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/11
Other Adverse Events (participants affected / at risk) | 0/3 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECP/Pent (N=3) | Pent (N=11)
ards (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
dvt (Vascular disorders) | 0 (0) | 3 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECP/Pent (N=3) | Pent (N=11)
skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No